CLINICAL TRIAL: NCT03604276
Title: Neuroinflammatory Response and Headache Control in Patients After Subarachnoid Hemorrhage (HASH4-CSF) - An Observational Trial
Brief Title: Neuroinflammatory Response and Headache Control in Patients After Subarachnoid Hemorrhage
Acronym: HASH4-CSF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Elizabeth Glisic, Clinical Pharmacist, MaineHealth
Other Study IDs: 1100316-599
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Headache; Subarachnoid Hemorrhage
Keywords: Headache; Subarachnoid hemorrhage; Neuroinflammation
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the relationship between the Neuroinflammatory response and headache pain after subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Persistent headache is a significant medical issue that affects 20% of patients who survive an aneurysmal subarachnoid hemorrhage (SAH). This headache may last years, severely affecting quality of life. Laboratory evidence suggests that the persistent headache may be a result of a maladaptive neuroinflammatory response to the hemorrhage injury that is more vigorous than necessary. The goal of this study is to measure key immunomodulators in the blood and the cerebrospinal fluid of these patients in order to determine the magnitude and dynamics of their neuroinflammatory response. In addition, the investigators will collect and analyze observational data about the success of medications to treat headache, with a specific focus on the anti-inflammatory agent dexamethasone, in managing acute headache pain and preventing the development of persistent headaches in patients after SAH.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic subarachnoid hemorrhage
* Age > 18 years
* Treated with external ventricular drainage

Exclusion Criteria:

* Pregnancy or lactation
* Age < 18 years
* Traumatic SAH

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible patients are patients with a non-traumatic subarachnoid hemorrhage who are treated with an external ventricular drain for symptomatic hydrocephalus.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the neuroinflammatory response in the CSF and blood of patients with non-traumatic SAH. | 10 days
Determination of correlation between the neuroinflammatory response and severity/presence of headache pain. | 10 days
Determination of correlation between the neuroinflammatory response and development of chronic headache. | 1 year

SECONDARY OUTCOMES:
Comparison of the neuroinflammatory response in the CSF and blood in patients treated with dexamethasone versus other analgesics post SAH. | 10 days
Comparison of dexamethasone versus other analgesics in their ability to improve measures of quality of life. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Glisic, PharmD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: Undecided